CLINICAL TRIAL: NCT04727788
Title: Validation of Genomic Immune-phenotyping Profiles in Peripheral Blood Gene Signatures to Predict Risk of Kidney Transplant Rejection
Brief Title: Validation of Genomic Immune-phenotyping Profiles to Predict Risk of Kidney Transplant Rejection
Status: Active, not recruiting | Type: Observational
Sponsor: Verici Dx (Industry)
Responsible Party: Sponsor
Other Study IDs: VDX 20-1001
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplant Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, urine, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Global, non-randomized, observational study for the validation of Verici Dx genomic tests to predict risk of kidney clinical and subclinical acute rejection, and chronic allograft damage or interstitial fibrosis / tubular atrophy by correlating peripheral blood gene expression profiles with graft injury (e.g. cellular / antibody-mediated), rejection and death censored graft loss.

DETAILED DESCRIPTION:
The study is correlative and observational and will involve collecting clinical and pathological data along with blood, biopsy tissue and urine during standard routine scheduled medical visits for transplant preparation or monitoring. The blood will be used for next generation sequencing in the Verici Dx laboratory to create transcriptomic profiles to validate performance characteristics of three Verici Dx sequencing immune-phenotype signature risk score tests. The research biopsy tissue and urine are for secondary or exploratory objectives. To allow comparison with current accepted standard approaches to identify kidney transplant injury or rejection, digital images of stained tissue sections taken from surveillance or for-cause biopsy tissue will be evaluated in a central pathology laboratory for the purposes of this study. Enrolled subjects will continue in the study for 24 months during which the planned validation of the acute clinical and subclinical rejection tests will complete after 6 months of follow-up; subjects will be followed to 24 months for the validation of the Verici Dx blood-based fibrosis risk prognostic test. After 24 months, patients will be followed through ANZDATA and UNOS registry data for later development of fibrosis or for graft loss or death.

ELIGIBILITY:
Inclusion Criteria:

1. Individual Recipients of living or deceased donor kidney transplant
2. Age: ≥ 18 ≤ 80
3. The subject must be able to comprehend and sign an approved informed consent form

Exclusion Criteria:

1. Recipients of multiple organ transplant, except kidney-pancreas multiple transplant
2. Subjects who are currently participating in a therapeutic clinical trial for transplant rejection
3. HIV or Hepatitis C positive patients
4. Persons who are known to be pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney or kidney/pancreas transplant patients
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2021-03-21 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pre-transplant: test for prediction of risk of Early Acute Rejection (EAR) | baseline
  early acute rejection occurring within first 6 months, including borderline ACR
Acute Cellular Rejection (ACR): test to identify the risk of clinical and sub-clinical ACR | 6 months
  clinical or subclinical acute rejection 3 months post transplant including borderline ACR, acute cell-mediated rejection as confirmed by histologic evidence on biopsy
Fibrosis: test to predict the risk of developing fibrosis of the allograft and allograft loss | 24 months
  clinical or subclinical acute rejection due to fibrosis 12 months post transplant as confirmed by histologic evidence on biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Donovan, PhD, MD, Principal Investigator — Verici Dx
Locations (13):
- United States (9):
  - University of Illinois at Chicago, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - University of Maryland, Baltimore, Maryland
  - Henry Ford, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Washington, Seattle, Washington
- CHU Grenoble Alpes Health Center, Grenoble, France
- Italy (2):
  - Bologna University, Bologna
  - Brescia University, Brescia
- University Hospital Vall d'Hebron, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No